CLINICAL TRIAL: NCT03688204
Title: Clinical Implementation of a Polygenic Risk Score (PRS) for Breast Cancer: Impact on Risk Estimates, Management Recommendations, Clinical Outcomes, and Patient Perception
Brief Title: Clinical Implementation of a Polygenic Risk Score (PRS) for Breast Cancer
Status: Completed | Type: Observational
Sponsor: Ambry Genetics (Industry)
Responsible Party: Sponsor
Other Study IDs: SNP-17-001
Record Dates: First submitted 2018-09-20; First posted 2018-09-28 (Actual); Last update posted 2022-03-07 (Actual); Status verified 2022-03

CONDITIONS: Breast Cancer Risk
Keywords: Breast Cancer; Breast Neoplasm; Genetic Testing; Breast Cancer Risk; Cancer Risk; Risk Score; Genetic Risk Score; Polygenic Risk Score; Personalized Risk Score
MeSH Terms: conditions — Breast Neoplasms; Genetic Risk Score

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Residual specimen may be maintained for an indefinite period of time at Ambry Genetics and be available for future studies as provided for in the consent document. Future studies on identifiable specimens or data will require review by an IRB or ethics committee.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study aims to assess how a polygenic risk score (PRS) reported with the results of multi-gene panel testing affects the breast cancer risk management recommendations healthcare providers make to their patients. The PRS is a score based on small genetic changes, clinical history, and family history. The PRS is used to estimate remaining lifetime risk of developing breast cancer for patients with no personal history of breast cancer and an overall negative result from MGPT.

ELIGIBILITY:
Inclusion Criteria:

* Female, age ≥ 18 years
* Willing and able to provide meaningful informed consent
* Willing and able to complete study procedures as described in this protocol
* Electing to undergo multi-gene panel testing for hereditary breast cancer for clinical purposes at the time of consent
* No personal history of cancer (except non-melanoma skin cancer) and meets NCCN guidelines for BRCA1/2 testing based on family history of breast and/or ovarian cancer
* Meets Ambry criteria for clinical reporting of PRS score

Exclusion Criteria:

* Prior germline BRCA1/2 testing
* Not willing to receive PRS
* Personal history of cancer, except non-melanoma skin cancer
* Personal history of allogenic bone marrow/stem cell transplant

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will include 2000 individuals with a family history of breast and/or ovarian cancer who present for genetic counseling at one of the investigative sites. The investigative sites will be clinics that regularly sees patients that meet the above description.
Sampling Method: Probability Sample
Enrollment: 118 (Actual)
Dates: Start 2018-09-21 (Actual); Primary Completion 2020-11-11 (Actual); Study Completion 2020-11-11 (Actual)

PRIMARY OUTCOMES:
Change in Breast Cancer Risk Management Recommendations | First recommendations will be made within 45 days of the initial study visit. Second recommendations will be made within 75 days of the initial study visit.
  Breast Cancer Risk Management Recommendations are recorded at two separate times; first recommendations will be recorded by the investigator or his/her designee based on the results of MGPT only. After these recommendations are recorded, the complete report including the PRS will be released. Then the healthcare provider will record recommendations again based on the results of MGPT and PRS. The difference between these recommendations will be used as a measure of the effect a PRS has on breast cancer risk management recommendations made by healthcare providers.

CONTACTS AND LOCATIONS:
Overall Officials: Brigette Tippin-Davis, PhD, Study Director — Ambry Genetics
Locations (3):
- United States (3):
  - Providence Roy and Patricia Disney Family Cancer Center, Burbank, California
  - St Joseph Hospital of Orange, Orange, California
  - Edwards Comprehensive Cancer Center, Huntington, West Virginia